CLINICAL TRIAL: NCT07268404
Title: A 12-Week Virtual, Randomized, Double-Blind, Placebo-Controlled Trial Evaluating the Effects of Daily Nouri Hormone Balance Probiotic on Metabolic, Inflammatory, and Symptom Outcomes in Women
Brief Title: Women's Hormonal and Metabolic Wellbeing Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Daily Nouri (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: DNO001_14865
Record Dates: First submitted 2025-11-17; First posted 2025-12-05 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-11

CONDITIONS: Metabolic Health
Keywords: dietary supplement; quality of life; women's health; hormone balance

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: Dietary Supplement Capsule (Experimental): Hormone Balance Probiotic blend
  Interventions: Dietary Supplement: Probiotic Blend Capsule
- Placebo: Capsule (Placebo Comparator): Identical capsule containing inactive ingredients
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic Blend Capsule — Hormone Balance Probiotic Blend
  Arms: Intervention: Dietary Supplement Capsule
Dietary Supplement: Placebo — Placebo
  Arms: Placebo: Capsule

SUMMARY:
The goal of this clinical trial is to learn if Daily Nouri Hormone Balance Probiotic blend can improve metabolic, inflammatory, and symptom outcomes in women.

Participants will:

* Take the probiotic blend or placebo every day for 12 weeks
* Complete virtual assessments and report symptoms throughout the study

DETAILED DESCRIPTION:
This study is a 12-week, prospective, randomized, controlled clinical trial. It is an interventional study with participants assigned to either an active or control group. All study visits will be conducted virtually, including completion of questionnaires, collection of blood samples, and other assessments.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported irregular menstrual cycles, defined as one or more of the following:

  * Cycle length typically >35 days OR <21 days
  * Fewer than 9 menstrual periods in the past year
  * Unpredictable cycle timing (varies by >7 days month-to-month)
  * Irregular cycles present for ≥6 months
* One or more of the following hormonal balance concerns: skin, unwanted hair growth, hair thinning, weight concerns)
* Self-reported emotional symptoms that fluctuate with menstrual cycle, including:

  * Mood swings or irritability
  * Feelings of stress or tension
  * Low mood or feeling down
  * Difficulty with emotional regulation
* Not currently using hormonal therapies, metformin, GLP-1 receptor agonists, or anti-androgens.
* If taking supplements for menstrual/hormonal support: willing to discontinue for 2-week washout before baseline
* Weight stable (+ 5 pounds) for the past 2 months, not planning to start a new diet, exercise program, or medications during study
* Able to provide electronic informed consent.
* Willing to complete online surveys and at-home DBS sample collection.
* Negative home pregnancy test at baseline.
* Access to a computer or smartphone and reliable internet connection.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — women
Enrollment: 60 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Women's Health Quality of Life Scores | From baseline to week 12
  Women's Health Quality of Life as measured by changes in total and domains scores on the Health-Related Quality of Life Questionnaire for Polycystic Ovary Syndrome-26 (PCOSQ-26). Response Scale: 7-Point Likert Scale Per-Item Range: minimum: 1, maximum: 7, where higher scores indicate better outcomes.

SECONDARY OUTCOMES:
Overall Health Quality of Life Scores | 12 weeks
  Assessed by monthly Patient-Reported Outcomes Measurement Information System - 29 Profile (PROMIS-29) questionnaire. 28 items use 5-point Likert scale responses (0-4), 1 item is a numeric rating scale (0-10). For negatively-worded concepts higher scores indicate worse outcomes, for positively-worded concepts higher scores indicate better outcomes.
Change from baseline to Week 12 in Fasting Blood Glucose | 12 weeks
  Fasting Blood Glucose will be analyzed from dried blood spots (DBS), reported as mg/dL (milligrams per deciliter).
Change from baseline to Week 12 in Glycated Hemoglobin A1c (HbA1c) | 12 weeks
  HbA1c will be analyzed from dried blood spots (DBS), reported as percentage (%).
Change from baseline to Week 12 in High-Sensitivity C-Reactive Protein (hsCRP). | 12 weeks
  hsCRP will be analyzed from dried blood spots (DBS), reported as mg/L (milligrams per liter).
Supplementary Question - Sleep | 12 weeks
  Over the past 7 days, how would you rate your sleep quality overall? Visual Analog Scale, (0 = very poor, 10 = excellent) Over the past 7 days, how would you rate your energy level? Visual Analog Scale (0 = no energy/extremely fatigued, 10 = full energy/not fatigued at all)
Supplementary Question - Acne Severity | 12 weeks
  How would you rate the severity of your acne over the past 7 days? Visual Analog Scale, (Response: 0-10 scale, where 0 = no acne and 10 = severe acne)
Supplementary Question - Acne | 12 weeks
  To what extent does your acne currently affect your quality of life? (Response: 5-point Likert, from 'not at all' to 'extremely')
Supplementary Question - Sexual Health | 12 weeks
  Over the past 7 days, how would you rate your overall sexual interest and satisfaction? Visual Analog Scale (0 = Very poor, 10 = Excellent)

CONTACTS AND LOCATIONS:
Locations (1):
- Alethios, Inc., San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No